CLINICAL TRIAL: NCT04295525
Title: PHoral: Effects of Carnosine Supplementation on Quantity/Quality of Oral Salivae in Healthy Volunteer and in Subjects Affected by Common Oral Pathologies.
Brief Title: Carnosine Supplementation on Quantity/Quality of Oral Salivae.
Acronym: PHoral
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Michele Ciulla, Co-Principal Investigator, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P0A.20.20
Record Dates: First submitted 2020-02-26; First posted 2020-03-04 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Oral Diseases
Keywords: dental erosions; caries; périodontopathies
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Controls subjects placebo (Placebo Comparator): Placebo mucoadhesive oral tablet
  Interventions: Dietary Supplement: placebo mucoadhesive oral tablet
- Controls subjects active Treatment (Experimental): AqualiefTM 400 mg mucoadhesive oral tablet
  Interventions: Dietary Supplement: 400 mg mucoadhesive oral tablet
- Diseased subjects placebo (Placebo Comparator): Placebo mucoadhesive oral tablet
  Interventions: Dietary Supplement: placebo mucoadhesive oral tablet
- Diseased subjects active Treatment (Experimental): AqualiefTM 400 mg mucoadhesive oral tablet
  Interventions: Dietary Supplement: 400 mg mucoadhesive oral tablet

INTERVENTIONS:
Dietary Supplement: 400 mg mucoadhesive oral tablet — AqualiefTM (Metis Healthcare s.r.l., Milano, Italy)
  Arms: Controls subjects active Treatment; Diseased subjects active Treatment
Dietary Supplement: placebo mucoadhesive oral tablet — placebo
  Arms: Controls subjects placebo; Diseased subjects placebo

SUMMARY:
The aim of this study is to elucidate the mutual relationship between salivae characteristics and oral microbiome and to compare them with common oral disease; furthermore, by using specific bioinformatic tools to analyse the data, the potentials of Carnosine in preventing/treating oral diseases and its mechanism of action will be addressed by using quantitative proteomics.

DETAILED DESCRIPTION:
The pH of the oral cavity is a synthetic parameter that underlies a multifactorial process of continuous adjustment that includes the effect of salivae as a buffer and the contribution of the oral cavity microbiome. In some diseases of the oral cavity an alteration of these adjustment mechanisms is supposed to alter the normal flow of salivae and, consequently, the pH and the oral microbiome with the expansion of potentially pathogenic strains such as e.g. streptococcus viridans.

Carnosine (Car) is an endogenous dipeptide, composed of β-alanine and L-histidine, that was originally discovered in larger amounts in skeletal muscle of some vertebrates, including humans, showing a greater dependence on non-oxidative forms of energy metabolism. This peculiar association with muscular tissue and its pH-buffering properties has led to associate Car with the intracellular acid-base homeostasis of muscles. More recently, the physiological role of Car has been expanded beyond the intracellular buffering properties, supporting a role in sarcoplasmic Ca2+ regulation and neutralisation of reactive oxygen species (ROS). It is well known that ROS induce the formation of reactive electrophilic carbonyl species by reacting with lipids and sugars which, in turn, react with proteins forming irreversible adducts (AGEs, ALEs and EAGLEs) and cross-links that may affect the cardiovascular wall matrix that becomes less distensible, especially during the ageing process and/or diseases. Thus it is thought that Car and, indeed, other histidine-containing peptide (HCD), may prevent chronic diseases via their anti-inflammatory, anti-oxidative, anti-glycating, anti-ischaemic and chelating properties. Furthermore, the localisation of Car in other tissues such as brain, olfactory bulb, heart, stomach, pancreas, kidney has suggested further potential uses in preventing e.g. neurodegenerative disorder and cognitive function or the development of type II diabetes.

The oral microbiome (OM) is a relevant part of the whole human MO since it contains several different niches, with distinct microbial communities, colonising the oral cavity (OC), including not only bacteria but also fungi, viruses, archaea and protozoa. These communities form a complex ecological system that influences OC and systemic health. Indeed the prevalent oral diseases (OD), namely dental caries and periodontal diseases, are believed to be microbiota-related. Furthermore, several evidences support the theory that many systemic diseases are associated with an altered OM, among these the most frequently associated diseases are metabolic, such as diabetes, cardiovascular and oncological ones. For their prevalence worldwide, among OD, periodontal infection, including gingivitis and chronic periodontitis, is possibly the most prevalent human microbial diseases (HMD).

In order to protect the OC from HMD, in the present project Car has been chosen as a possible preventive and/or therapeutic principle for its aforementioned multiple biological effects. Thus the safety and efficacy of AqualiefTM (Metis Healthcare s.r.l., Milano, Italy) a 400 mg mucoadhesive oral tablet (13 x 4 mm), that recognise Car as main ingredient, will be tested on healthy volunteer and in subjects affected by common OD.

The main objectives of this protocol are to estimate the quantity/quality of oral salivae and OM in healthy volunteer and in patients affected by common OD, before and after 7 days of treatment with AqualiefTM, 1 tablet twice. The characteristics of oral salivae (Sal) that will be studied are:

a - unstimulated and stimulated (paraffin-activated) salivary flow rates, pH and buffering power; b - quantitative proteomics (QP), on selected targets, representing the main metabolites/components of OM.

By matching Sal characteristics with OM and comparing them with OD, it is expected to elucidate their mutual relationship; furthermore, by using specific bioinformatic tools to analyse the data, the potentials of Car in preventing/treating OD and its mechanism of action will be addressed by using QP.

The study will take place at the Odontoiatric University Clinic (OUC), Istituto Stomatologico Italiano (ISI) of Milan, Italy, in a prospective, randomised, double-blind, placebo-controlled fashion.

ELIGIBILITY:
Inclusion Criteria for Oral Diseased subjects:

* dental erosions (De)
* caries (Ca)
* périodontopathies (Pe)

Exclusion Criteria for both:

* allergies/intolerances to the consumption of Carnosine
* taking other food supplements
* any type of drug treatment (interview)
* smoking
* pregnancy/lactation
* any systemic diseases such as cardiovascular and respiratory, diabetes mellitus, HIV infection, or inflammatory conditions causing non-plaque dependent OD.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Effects on oral pH. | 7 days
  Any change of oral pH from basal.
Saliva Production unstimulated. | 7 days
  Change of oral saliva production, unstimulated.
Saliva Production stimulated. | 7 days
  Change of oral saliva production, stimulated.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Ciulla, MD, Principal Investigator — Lab. Clin. Informatics & Cardiovascular Imaging, University of Milan
Locations (1):
- Department of Biomedical, Surgical, and Dental Sciences, Istituto Stomatologico Italiano, Aesthetic Dentistry, School of Dentistry, University of Milan, Milan, Italy., Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Almeida Pdel V, Gregio AM, Machado MA, de Lima AA, Azevedo LR. Saliva composition and functions: a comprehensive review. J Contemp Dent Pract. 2008 Mar 1;9(3):72-80. PMID 18335122
- [Result] Marsh PD, Do T, Beighton D, Devine DA. Influence of saliva on the oral microbiota. Periodontol 2000. 2016 Feb;70(1):80-92. doi: 10.1111/prd.12098. PMID 26662484
- [Result] Grassl N, Kulak NA, Pichler G, Geyer PE, Jung J, Schubert S, Sinitcyn P, Cox J, Mann M. Ultra-deep and quantitative saliva proteome reveals dynamics of the oral microbiome. Genome Med. 2016 Apr 21;8(1):44. doi: 10.1186/s13073-016-0293-0. PMID 27102203
- [Result] Abranches J, Zeng L, Kajfasz JK, Palmer SR, Chakraborty B, Wen ZT, Richards VP, Brady LJ, Lemos JA. Biology of Oral Streptococci. Microbiol Spectr. 2018 Oct;6(5):10.1128/microbiolspec.gpp3-0042-2018. doi: 10.1128/microbiolspec.GPP3-0042-2018. PMID 30338752
- [Result] Dolan E, Saunders B, Harris RC, Bicudo JEPW, Bishop DJ, Sale C, Gualano B. Comparative physiology investigations support a role for histidine-containing dipeptides in intracellular acid-base regulation of skeletal muscle. Comp Biochem Physiol A Mol Integr Physiol. 2019 Aug;234:77-86. doi: 10.1016/j.cbpa.2019.04.017. Epub 2019 Apr 25. PMID 31029715
- [Result] Boldyrev AA, Aldini G, Derave W. Physiology and pathophysiology of carnosine. Physiol Rev. 2013 Oct;93(4):1803-45. doi: 10.1152/physrev.00039.2012. PMID 24137022
- [Result] Ciulla MM, Paliotti R, Carini M, Magrini F, Aldini G. Fibrosis, Enzymatic and Non-Enzymatic Cross-Links in Hypertensive Heart Disease. Cardiovasc Hematol Disord Drug Targets. 2011;11(2):61-73. doi: 10.2174/187152911798347025. PMID 22044034
- [Result] Menon K, Mousa A, de Courten B. Effects of supplementation with carnosine and other histidine-containing dipeptides on chronic disease risk factors and outcomes: protocol for a systematic review of randomised controlled trials. BMJ Open. 2018 Mar 22;8(3):e020623. doi: 10.1136/bmjopen-2017-020623. PMID 29567852
- [Result] Zhang Y, Wang X, Li H, Ni C, Du Z, Yan F. Human oral microbiota and its modulation for oral health. Biomed Pharmacother. 2018 Mar;99:883-893. doi: 10.1016/j.biopha.2018.01.146. Epub 2018 Feb 20. PMID 29710488
- [Result] Holtfreter B, Albandar JM, Dietrich T, Dye BA, Eaton KA, Eke PI, Papapanou PN, Kocher T; Joint EU/USA Periodontal Epidemiology Working Group. Standards for reporting chronic periodontitis prevalence and severity in epidemiologic studies: Proposed standards from the Joint EU/USA Periodontal Epidemiology Working Group. J Clin Periodontol. 2015 May;42(5):407-12. doi: 10.1111/jcpe.12392. Epub 2015 May 7. PMID 25808877